CLINICAL TRIAL: NCT01642940
Title: Τicagrelor Versus Prasugrel in Diabetic Patients: a Pharmacodynamic Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor of Cardiology, Director of Cardiology Department, University of Patras
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-11
Record Dates: First submitted 2012-07-12; First posted 2012-07-17 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prasugrel (Active Comparator)
  Interventions: Drug: Prasugrel
- Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor

INTERVENTIONS:
Drug: Prasugrel — Prasugrel 10mg/day
  Arms: Prasugrel
Drug: Ticagrelor — Ticagrelor 90mg twice a day
  Arms: Ticagrelor

SUMMARY:
This is a prospective, randomized, single-center, single blind, investigator initiated, two period study of crossover design. Diabetic patients with Acute Coronary Syndrome (ACS), treated with oral and/or parenteral hypoglycaemic therapy for at least 1 month and subjected to percutaneous coronary intervention (PCI), will be randomized after a baseline platelet reactivity (PR) assessment (24 hours post PCI) while under clopidogrel in a 1:1 ratio to either prasugrel 10mg or ticagrelor 180mg for 15 days followed by crossover directly to the alternate therapy for an additional 15 days without an intervening washout period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years
* Diabetic patients treated with oral and/or parenteral hypoglycaemic therapy for at least 1 month
* Patients with acute coronary syndrome subjected to PCI with a baseline PR evaluation 24 hours post PCI while on clopidogrel
* Informed consent obtained in writing

Exclusion Criteria:

* Treatment with other investigational agents (including placebo) or devices within 30 days prior to randomization or planned use of investigational agents or devices prior to the Day 30 visit.
* Pregnancy
* Breastfeeding
* Inability to give informed consent or high likelihood of being unavailable for the Day 30 follow up.
* Cardiogenic shock
* Major periprocedural complications (death, stent thrombosis, vessel perforation, arrhythmias requiring cardioversion, temporary pacemaker insertion or intravenous antiarrhythmic agents, respiratory failure requiring intubation, vascular injury (pseudoaneurysm, arteriovenous shunt, retroperitoneal bleeding or hematoma >5 cm at the arterial catheter insertion site), major bleeding (need for bood transfusion or drop in haemoglobin post-PCI by ≥ 5 gr/ dl or intracranial bleeding).
* Unsuccessful PCI (residual stenosis > 30% or flow < ΤΙΜΙ 3) or planned staged PCI in the next 30 days after randomization
* Requirement for oral anticoagulant prior to the Day 30 visit
* Current or planned therapy with other thienopyridine class of ADP receptor inhibitors.
* Known hypersensitivity to prasugrel or ticagrelor
* History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 6 months.
* Other bleeding diathesis, or considered by investigator to be at high risk for bleeding on longterm thienopyridine therapy.
* Any previous history of ischemic stroke, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm).
* Thrombocytopenia (< 100.000/μL) at randomization
* Anaemia (Hct < 30%) at randomization
* Polycytaemia (Hct > 52%) at randomization
* Periprocedural IIb/IIIa inhibitors administration
* Severe allergy to contrast agent, unfractionated heparin, enoxaparin or bivalirudin that cannot be adequately premedicated.
* Recent (< 6 weeks) major surgery or trauma, including GABG.
* Subjects receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors that cannot be discontinued for the duration of the study.
* Concomitant oral or IV therapy with strong CY P3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazana vir, grapefruit juice N1 L/d), CYP3A substrates with narrow therapeutic indices (cyclosporine, quinidine), or strong CYP3A inducers (rifampin /rifampicin, phenytoin, carbamazepine).
* Increased risk of bradycardiac events.
* Dialysis required.
* Age ≥ 75 years
* Weight < 60 Kg
* Severe hepatic impairment
* Severe uncontrolled chronic obstructive pulmonary disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | 15 days
  The primary outcome will be assessed 15 days after the onset of each study drug by the VerifyNow (Accumetrics)assay in platelet reactivity units (PRU)

SECONDARY OUTCOMES:
Hyporesponsiveness rate (PRU≥230) at the end of the 2 treatment periods | Day 15
  Hyporesponsiveness rate will be assessed 15 days after the onset of each study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department Patras University Hospital, Pátrai, Achaia, Greece

REFERENCES:
- [Derived] Alexopoulos D, Xanthopoulou I, Mavronasiou E, Stavrou K, Siapika A, Tsoni E, Davlouros P. Randomized assessment of ticagrelor versus prasugrel antiplatelet effects in patients with diabetes. Diabetes Care. 2013 Aug;36(8):2211-6. doi: 10.2337/dc12-2510. Epub 2013 Mar 14. PMID 23491524